CLINICAL TRIAL: NCT07347236
Title: MyNOURISH: Effectiveness of Hydrolysed Collagen on Nutritional, Functional, Body Composition and Bone Health Among Older Adults With Fragility Fractures in Hospital Sultan Abdul Aziz. .
Brief Title: MyNOURISH: Hydrolysed Collagen Supplementation in Older Adults With Fragility Fractures
Acronym: MyNOURISH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Pengajar Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MyNOURISH2025
Record Dates: First submitted 2025-12-21; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Fragility Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Hydrolysed Collagen supplement) (Experimental): Participants in this group will receive 15 g of hydrolysed tilapia collagen (PROTÉGEN Plus) daily for 12 weeks. Participants will attend follow-up assessments at baseline, week 6, week 12, and week 24 to monitor adherence, safety, and outcomes. Unopened supplement sachets will be returned at week 6 and 12 to assess compliance.
  Interventions: Dietary Supplement: Hydrolysed Collagen (PROTÉGEN Plus)
- Control Group (Standard Multidisciplinary Care) (Active Comparator): Participants receive standard multidisciplinary care without collagen supplementation.
  Interventions: Other: Standard Multidisciplinary Care

INTERVENTIONS:
Dietary Supplement: Hydrolysed Collagen (PROTÉGEN Plus) — Participants will receive 15 g of hydrolysed tilapia collagen (PROTÉGEN Plus) daily for 12 weeks, in addition to usual care provided within a multidisciplinary team approach.
  Arms: Intervention Group (Hydrolysed Collagen supplement)
Other: Standard Multidisciplinary Care — Usual care consists of routine medical, nutritional, and rehabilitation management delivered through a multidisciplinary team approach at HSAAS, including follow-up medical reviews by physicians, personalised dietary counselling by dietitians, and tailored rehabilitation sessions conducted by physiotherapists.
  Arms: Control Group (Standard Multidisciplinary Care)

SUMMARY:
The goal of this clinical trial is to learn whether hydrolysed collagen supplementation (PROTÉGEN Plus) within multidisciplinary care can improve nutrition and recovery in older adults with fragility fractures.

The main questions this study aims to answer are:

1. Does collagen supplementation improve malnutrition status, nutritional biomarker (albumin levels), body composition (skeletal muscle and fat-free mass), functional capacity and bone turnover (P1NP and CTX) over 12 weeks intervention period?
2. Does hydrolysed collagen supplementation have additional effects on the malnutrition status and functional capacity among older adult outpatients with fragility fractures at Week 6?
3. Are the effects of hydrolysed collagen supplementation on the malnutrition status, nutritional biomarker (albumin), body composition (skeletal muscle and fat-free mass), functional capacity, and bone turnover biomarkers (P1NP and CTX) sustained up to 24 weeks post-intervention compared to standard care?

Researchers will compare two groups of older adults (aged 60 years and above) receiving care at Hospital Sultan Abdul Aziz Shah (HSAAS), Universiti Putra Malaysia:

- Intervention group: Participants will receive hydrolysed collagen (PROTÉGEN Plus) with usual care within a multidisciplinary team for 12 weeks.

Attend study visits at baseline, week 6, week 12, and week 24 (for follow-up of sustained effects). Keep a diary to record supplement intake, adherence, and any side effects, and return unopened supplement sachets at week 6 and 12 to monitor compliance.

- Control group: Participants will receive usual care within a multidisciplinary team. Attend study visits at baseline, week 6, week 12, and week 24 (for follow-up of sustained effects).

This study will help researchers understand whether adding tilapia-derived collagen supplementation to multidisciplinary care can support better nutrition, muscle and bone health, and long-term recovery in older adults after a fragility fracture. It is hoped that the findings will strengthen the evidence for incorporating targeted nutritional strategies as part of fragility fracture management and secondary fracture prevention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 60 years and above.
* History of a fragility fracture (e.g., hip, wrist, or vertebral fracture) sustained within the past 12 months.
* Registered outpatient at Hospital Sultan Abdul Aziz Shah (HSAAS).
* Malaysian citizen.
* Able to communicate in Bahasa Malaysia or English.
* Able and willing to provide written informed consent.
* Cognitive function score >4 on the Elderly Cognitive Assessment Questionnaire (ECAQ).
* Currently undergoing a structured rehabilitation programme.
* May be receiving antiresorptive osteoporosis therapy or not receiving any osteoporosis pharmacological treatment at the time of recruitment.

Exclusion Criteria:

* Cognitive impairment, defined as ECAQ score ≤4
* Metabolic bone diseases other than osteoporosis (e.g., Paget's disease, osteomalacia).
* Severe endocrine or metabolic disorders affecting bone metabolism (e.g., primary hyperparathyroidism, Cushing's syndrome, hyperthyroidism, hypogonadism, acromegaly).
* Terminal illness or palliative care needs (e.g., advanced cancer, end-stage organ failure, late-stage neurodegenerative diseases).
* Known allergy to fish, seafood, or collagen supplements, or diagnosis of phenylketonuria.
* Kidney disease, including history of kidney stones or chronic kidney disease stage 4-5 (estimated glomerular filtration rate <44 mL/min/1.73 m²).
* Participation in another interventional study that may interfere with the study protocol.
* Use of nutritional supplements during the study period.
* Prior use of collagen or amino acid-based supplements within the past 6 months.
* Non-ambulatory status prior to the fracture.
* Unstable medical conditions (e.g., uncontrolled arrhythmias, recent myocardial infarction, unstable angina, uncontrolled hypertension, pulmonary embolism).
* Current use of anabolic osteoporosis therapy.
* Alcohol dependence or active alcoholism.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Malnutrition status | Baseline, Week 6, Week 12, and Week 24 (follow-up for sustainability of effects)
  Malnutrition status will be assessed using the Mini Nutritional Assessment-Short Form (MNA-SF). The score categorizes participants as well-nourished, at risk of malnutrition, or malnourished. The study will evaluate the improvement in malnutrition status through the scoring on each timepoints, following hydrolysed collagen supplementation compared with standard multidisciplinary care.

SECONDARY OUTCOMES:
Nutritional Biomarker (Serum albumin level) | Baseline, Week 12, and Week 24 (follow-up for sustainability of effects)
  Serum albumin concentration will be measured from fasting blood samples to assess improvement in nutritional biomarker status. Increased albumin levels indicate improved protein status following hydrolysed collagen supplementation compared with standard multidisciplinary care.
Body composition (skeletal muscle mass and fat-free mass) | Baseline, Week 12, and Week 24 (follow-up for sustainability of effects)
  Body composition-including skeletal muscle mass and fat-free mass-will be measured using bioelectrical impedance analysis (BIA). Changes will reflect improvement in overall muscle and bone tissue composition among older adults receiving hydrolysed collagen supplementation compared with standard multidisciplinary care.
Functional capacity-Change in Short Physical Performance Battery (SPPB) score | Baseline, Week 6, Week 12, and Week 24 (follow-up for sustainability of effects)
  Functional capacity will be assessed using the Short Physical Performance Battery (SPPB). These measures evaluate lower-extremity performance, balance, gait speed, and upper-body strength, collectively reflecting participants' physical function and rehabilitation progress. The SPPB consists of three components: balance tests, gait speed, and repeated chair stands. Scores range from 0 to 12, with higher scores indicating better physical performance. Improvements in these outcomes will be used to determine the added effect of hydrolysed collagen supplementation compared with standard multidisciplinary care alone.
bone turnover biomarkers - Change in serum procollagen type I N-terminal propeptide (P1NP) levels | Baseline, Week 12, and Week 24 (follow-up for sustainability of effects)
  Serum procollagen type I N-terminal propeptide (P1NP) will be measured as a marker of bone formation. Changes in P1NP levels reflect the bone synthesis. Improvements indicate enhanced bone metabolism following hydrolysed collagen supplementation compared with standard multidisciplinary care
Functional capacity - Change in handgrip strength | Baseline, Week 6, Week 12, and Week 24 (follow-up for sustainability of effects)
  Handgrip strength will be assessed using a hand-held dynamometer as a measure of muscle strength. Measurements will be obtained from the dominant hand, with the average of three trials recorded. Higher values indicate greater muscle strength. Units of measure is in Kilogram (Kg)
Bone Turnover Biomarker - Change in serum C-terminal telopeptide of type I collagen (CTX) levels | Baseline, Week 12, and Week 24
  Serum C-terminal telopeptide of type I collagen (CTX) will be measured as a biochemical marker of bone resorption. Changes in CTX reflect alterations in bone resorption following hydrolysed collagen supplementation compared with standard multidisciplinary care.

CONTACTS AND LOCATIONS:
Overall Officials: Noraida Omar, BSc(Dietetics), Ph.D(Nutrition, Principal Investigator — Department of Dietetics, Faculty of Medicine and Health Sciences, Universiti Putra Malaysia (UPM)
Locations (1):
- Hospital Sultan Abdul Aziz Shah (HSAAS), Universiti Putra Malaysia, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://hsaas.upm.edu.my/